CLINICAL TRIAL: NCT05854186
Title: Georgia: Technology and WIC - A Comprehensive Approach to Public Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Georgia Department of Public Health, Division of Health Promotion (Unknown); RTI International (Other)
Responsible Party: Principal Investigator, Erin Hennessy, Assistant Professor, Division of Nutrition Interventions, Communication and Behavior Change Director ad interim, ChildObesity180 Friedman School of Nutrition Science and Policy, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 211203
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Telehealth; Nutrition Education; Breast Feeding; Dietary Intake; WIC
Keywords: Telehealth; WIC; nutrition education; breast feeding; dietary intake
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Study participants will be clients at local WIC agency sites where either the telehealth solution is offered or where only usual care is available (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth solution (Experimental): Telehealth solution offered.
  Interventions: Behavioral: Telehealth solution: video conferencing
- Control (No Intervention): Usual care.

INTERVENTIONS:
Behavioral: Telehealth solution: video conferencing — Telehealth solution: video conferencing
  Arms: Telehealth solution

SUMMARY:
With funding through USDA and Tufts University's Telehealth Intervention Strategies for WIC (THIS-WIC) project, the Georgia WIC department will be implementing a telehealth solution for nutrition and breastfeeding support. The purpose of this study is to evaluate this telehealth solution. The research/evaluation involves completing online surveys. The evaluation will focus on participant satisfaction, usage of the telehealth solution, and use of information collected on the WIC participant through the WIC management information system (MIS). It is hypothesized that the telehealth solution will increase WIC participant's satisfaction with nutrition and breastfeeding support while also reducing the burden of attending in-person care.

DETAILED DESCRIPTION:
Telehealth can reduce barriers and increase access to care, and it can be applied to the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). WIC is a federal nutrition assistance program that helps low-income women with children up to age 5. There is a large volume of research that supports remote patient monitoring, and the most benefits are found when telehealth is used for communication and counseling. The USDA awarded Tufts University a grant to test and evaluate the use of telehealth innovations in the delivery of USDA's WIC program. Tufts University then offered the USDA/Tufts Telehealth Intervention Strategies for WIC (THIS-WIC) grant opportunity to WIC state agencies across the US. THIS-WIC selected 7 WIC State Agencies to receive grants, and the GA state agency is one recipient. The THIS-WIC team at Tufts University is leading the evaluation of these telehealth solutions in collaboration with funded WIC State Agencies.

THIS-WIC aims to generate evidence from GA's video-conferencing telehealth solution to inform how the telehealth platform supports WIC services compared to usual in-person care. Evaluation findings will inform stakeholders about the platform's benefits and how viable it is to sustain and adapt more widely.

The purpose of this study is to evaluate the effectiveness of this telehealth solution by having clients complete surveys on their comfortability using telehealth and their satisfaction with the telehealth appointment. Additionally, secondary demographic and other nutrition-related information about study participants is already collected in the MIS and will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Breastfeeding women
* postpartum women with children in the age range of 0 to 5 years

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2566 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the telehealth solution | During the study period, approximately 18 months
  WIC clients satisfaction with nutrition education and breastfeeding support offered via the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

SECONDARY OUTCOMES:
Breastfeeding duration | During the study period, approximately 18 months
  Duration of breastfeeding in clients offered the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants
Attendance at scheduled appointments | During the study period, approximately 18 months
  WIC clients attendance at appointments when offered the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Dietary intake | During the study period, approximately 18 months
  Impact of the telehealth solution compared to usual care on dietary intake. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Attitudes to breastfeeding and nutrition education | During the study period, approximately 18 months
  Impact of the telehealth solution compared to usual care on WIC clients' attitudes to breastfeeding and nutrition education. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Barriers encountered in obtaining nutrition education and breastfeeding support | During the study period, approximately 18 months
  Impact of the telehealth solution compared to usual care on barriers encountered by WIC clients in obtaining nutrition education and breastfeeding support. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hennessy, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No